CLINICAL TRIAL: NCT00519818
Title: A Phase 2, Open Label, Crossover Pharmacokinetic and Pharmacodynamic Study to Compare Chronocort Versus Cortef in Patients With CAH
Brief Title: Comparison of Two Forms of Hydrocortisone in Patients With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070211
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Congenital Adrenal Hyperplasia; 21-Hydroxylase Deficiency; Adrenogenital Syndrome
Keywords: Congenital Adrenal Hyperplasia; Hydrocortisone; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency; Adrenogenital Syndrome | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cortef and Chronocort (Experimental): Cortef 3 times daily(total dose 30 mg)for minimum of 7 days followed by Chronocort 30 mg once daily nigh time dose for 28 +/- 3 days duration
  Interventions: Drug: Chronocort; Drug: Cortef

INTERVENTIONS:
Drug: Chronocort — Chronocort 30 mg once daily nigh time dose for 28 +/- 3 days duration
  Other Names: Hydrocortisone modified release tablet treatment
Drug: Cortef — Cortef 3 times daily(total dose 30 mg)for minimum of 7 days
  Other Names: Hydrocortisone immediate release tablet

SUMMARY:
This study will test a new, extended release form of hydrocortisone called Chronocort in patients with congenital adrenal hyperplasia (CAH). People with CAH do not make enough of the adrenal hormones cortisol and aldosterone, and their adrenal glands make too much of the sex hormone androgen. Medicines called glucocorticoids (hydrocortisone, dexamethasone and prednisone) are currently used to treat CAH, but finding the best dose of these drugs that effectively lowers androgens without causing undesirable side effects, such as weight gain and slow growth rate in children, is often difficult to achieve.

Adolescents and adults with CAH due to 21-hydroxylase deficiency may be eligible for this study. Children 16 years of age and older are eligible with confirmation by bone age that they are no longer growing.

Participants undergo the following tests and procedures during two inpatient visits one month apart at the NIH Clinical Center:

* Medical history and physical examination.
* Medications: Following 7 days of Cortef (standard drug treatment for CAH), patients begin taking Chronocort on day 3 of hospitalization and continue the tablets once a day for 1 month.
* Blood tests: A catheter (plastic tube) is inserted in a vein and left in place for frequent blood draws in order to avoid repeated needlesticks. Blood is drawn for chemistries, blood count, pregnancy test in women, and for serial tests (up to 26 samples in a 24-hour period) to measure hormone levels.
* 24-hour urine test.
* Height and weight measurements.

Between the two hospitalizations, patients are contacted by NIH weekly to check for possible side effects from Chronocort. Two weeks after the first visit, patients also will have blood drawn by their regular doctor or a local clinic. A few days before the second hospitalization, patients undergo a 20-minute telephone questionnaire about energy level and well being.

About 30 days after discharge from the second hospitalization, patients are followed up with a telephone call to see how they are doing.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency is a disease of the adrenal cortex characterized by cortisol deficiency with or without aldosterone deficiency, and androgen excess. The severe or classic form occurs in 1 in 15,000 births worldwide, while the mild non-classic form is a common cause of hyperandrogenism. The discovery of glucocorticoid therapy as a treatment for CAH occurred in the 1950's resulting in patients with classic CAH surviving to live a normal lifespan. However, existing treatment is suboptimal and many unresolved clinical problems exist. Standard hormone replacement often fails to normalize the growth and development of children with CAH, and adults may experience iatrogenic Cushing syndrome, hyperandrogenism, infertility or the development of the metabolic syndrome. Chronocort, a newly-developed formulation of hydrocortisone, results in a slow release of hydrocortisone that is designed to mimic the normal cortisol circadian rhythm. This new medical strategy, physiologic cortisol replacement, offers the prospect of an improved outcome of treatment. Chronocort has been safely given to healthy adult males in pharmacokinetic studies. This first ever study in patients with CAH is a pharmacokinetic/pharmacodynamic study comparing Chronocort to Cortef, the conventional immediate-release form of hydrocortisone.

ELIGIBILITY:
* INCLUSION CRITERIA:

Satisfactory pre-trial screening

Provision of signed written informed consent and written assent from patients less than 18 years old, as applicable.

Good general health.

Females of childbearing potential must have a negative pregnancy test initially and at all visits. Females who are engaging in sexual intercourse must be using medically acceptable method of contraception.

EXCLUSION CRITERIA:

Co-morbid condition requiring daily administration of a medication that induces hepatic enzymes or interferes with the metabolism of glucocorticoids.

Clinical or biochemical evidence of hepatic or renal disease. Creatinine above the normal range or elevated liver function tests (Transaminases greater than 1.5 the upper limits of normal).

Females who are pregnant or lactating.

Patients with any other significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the trial.

Participation in another clinical trial of an investigational or licensed drug or device within 3 months prior to inclusion in this study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Merck, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Therrell BL. Newborn screening for congenital adrenal hyperplasia. Endocrinol Metab Clin North Am. 2001 Mar;30(1):15-30. doi: 10.1016/s0889-8529(08)70017-3. PMID 11344933
- [Background] Merke DP, Bornstein SR. Congenital adrenal hyperplasia. Lancet. 2005 Jun 18-24;365(9477):2125-36. doi: 10.1016/S0140-6736(05)66736-0. PMID 15964450
- [Background] Krieger DT, Allen W, Rizzo F, Krieger HP. Characterization of the normal temporal pattern of plasma corticosteroid levels. J Clin Endocrinol Metab. 1971 Feb;32(2):266-84. doi: 10.1210/jcem-32-2-266. No abstract available. PMID 4321505

RESULTS

PARTICIPANT FLOW:
Groups:
- Cortef Then Chronocort: Hydrocortisone immediate release tablet treatment then Modified release hydrocortisone
Period: Overall Study
Arm/Group | Cortef Then Chronocort
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cortef Then Chronocort: Hydrocortisone immediate release 3 times daily total dose 30mg for 7 days, then hydrocortisone modified release tablet 30mg once nightly for 28days
Arm/Group | Cortef Then Chronocort
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Chronocort vs. Cortef Cortisol Concentrations (AUC Over 24 Hours - Time Points 0,.5,1,1.5,2,3,4,5,6,7,8,10,10.5,11, 11.5,12,13,15,17,17.5,18,18.5,19,20,22,24 Post Dose).
Time Frame: Cortef after one week, Chronocort after one month
Population: Per protocol
Measure: Mean (Standard Error); unit: h*nmol/l
Groups:
- Cortef: Hydrocortisone immediate release tablet
- Chronocort: Hydrocortisone modified release tablet treatment
Arm/Group | Cortef | Chronocort
Number analyzed (Participants) | 14 | 14
h*nmol/l | 5380 (414) | 3973 (166)

2. Secondary Outcome: 17 Hydroxyprogesterone at 08.00 Hours
Time Frame: Cortef after one week compared with Chronocort after one month
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Cortef | Chronocort
Number analyzed (Participants) | 14 | 14
nmol/l | 16.4 (27.9) | 86.9 (181.7)

ADVERSE EVENTS:
Time Frame: Adverse events for each subject were followed for 1 week in Cortef, 4 weeks on Chronocort and 4 weeks follow-up.
Groups:
- Chronocort: Hydrocortisone modified release tablet
Arm/Group | Chronocort | Cortef
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronocort (N=14) | Cortef (N=14)
Headache (Nervous system disorders) | 4 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No